CLINICAL TRIAL: NCT06593574
Title: A Multicenter, Randomized, Blind Evaluation, Parallel-controlled, Superiority Clinical Trial of Spinal Robot System for Safety and Efficacy Evaluation of Assisted Laminectomy
Brief Title: Safety and Effectiveness Evaluation of Spinal Laminectomy Robot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: The Third Affiliated Hospital of Southern Medical University (Other Government); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D2024096
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: Lumbar Spinal Stenosis; Lumbar Disc Herniation
Keywords: Spinal robot; Laminectomy
MeSH Terms: conditions — Spinal Stenosis; Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robotic laminectomy group (Experimental): The laminectomy is performed with the assistance of a robot
  Interventions: Procedure: Robotic laminectomy
- Manual laminectomy group (Active Comparator): The laminectomy is performed by the surgeon without the assistance of a robot
  Interventions: Procedure: Traditional laminectomy

INTERVENTIONS:
Procedure: Robotic laminectomy — Surgical robots are used to assist with laminectomy
  Arms: Robotic laminectomy group
Procedure: Traditional laminectomy — Instead of relying on a surgical robot, doctors perform the laminectomy themselves with an ultrasonic osteotome
  Arms: Manual laminectomy group

SUMMARY:
The purpose of this clinical trial is to evaluate the effectiveness and safety of this spinal robot in assisting doctors to perform laminectomy in spinal surgery under the premise of ensuring the safety of the subjects and ensuring the scientific nature of the clinical trial.

DETAILED DESCRIPTION:
This is a multicenter, randomized, blind evaluation, parallel-controlled, and superiority clinical trial. The objective of this study is to evaluate the effectiveness and safety of a spinal robot in assisting surgeons in laminectomy. The experiment included 3 centers with a total sample size of 70. The experimental group is the robot laminectomy group (RL group), and the control group is the manual laminectomy group (ML group). Laminectomy in the RL group is performed robotically, while laminectomy in the ML group is performed by the physician using an ultrasonic osteotome. The primary outcome measure is the accuracy of laminectomy. Secondary outcome measures included JOA score, VAS score, laminectomy success rate, laminectomy time per spinal segment, total laminectomy time, operative time, amount of surgical bleeding, number of X-ray exposures and total dose, and planned area excision rate. The evaluation was completed by comparing the outcomes between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years old (including 18 and 80 years old), regardless of gender;
* Patients with complete clinical data, willing and able to sign informed consent;
* Patients with lumbar disc herniation, lumbar spinal stenosis, lumbar instability, lumbar spondylolisthesis, and lumbar fracture meet the indications for spinal laminectomy and undergoing open surgery；
* Patients with lumbar disc herniation, lumbar spinal stenosis, or lumbar instability have one of the following:

  1. It was not effective after 3 months of conservative treatment
  2. Symptoms seriously affect the quality of life
  3. cauda equina nerve injury
* Lumbar spondylolisthesis occurs in one of the following:

  1. Symptoms of II° and below slip were not relieved by non-surgical treatment
  2. Lumbar spondylolisthesis III° and above
  3. Symptoms of lumbar spinal stenosis
* The TLISS score of lumbar spine fracture is greater than or equal to 4 points.

Exclusion Criteria:

* Patients who are not suitable for robot-assisted surgery;
* Patients with existing implants in or near the vertebral body of the lesion;
* Patients whose vertebral lamina bone tissue of the focal vertebra or adjacent vertebra has been removed;
* Pregnant and lactating female patients;
* the subject is unwilling or unable to restrict activities or follow medical advice;
* Patients with infection near the focal area;
* The patient is mentally incapable or unable to understand the requirements for participating in the study;
* The patient is critically ill, the expected survival period is not more than 2 years, and it is difficult to make an accurate assessment of the effectiveness and safety of the device;
* Patients with coagulation dysfunction;
* Other researchers did not consider it suitable for admission.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy rate of laminectomy | Immediately after the intraoperative laminectomy procedure
  According to the classification criteria for the accuracy of laminectomy proposed by Zhuofu Li, grade A indicates that the pre-planned cutting lines are basically located in the actual cutting groove or that the maximum distance between them is <1mm; Grade B indicates that the maximum distance between the pre-planned cutting line and the actual cutting groove is 1 to 2mm. Grade C indicates a maximum distance of >2 mm between the two. Grades A and B are acceptable. The percentage of A+B in the total number of planned boundaries was counted as the accuracy rate of laminectomy.

SECONDARY OUTCOMES:
Success rate of laminectomy | Immediately after the intraoperative laminectomy procedure
  After the laminectomy is complete, check whether the laminectomy can be successfully removed. Each cutting plane is evaluated individually.
Improvement rate of Japanese Orthopaedic Society (JOA) Score | JOA scores were used to evaluate experimental and control subjects before and one month after surgery.
  The JOA score is a scoring system used to assess lumbar dysfunction. The lumbar JOA score includes subjective symptoms (9), clinical signs (6), limits of daily activities (14), and bladder function (-6 to 0) on a 29-point scale. The lower the score, the more significant the dysfunction.
  Improvement rate = [(post-treatment score - pre-treatment score)/(29 - pre-treatment score)] × 100%.
Visual analogue scale (VAS) | Before and one month after the operation
  Visual analog scale, which indicates the degree of pain. The VAS score was used to evaluate the pain degree of the experimental group and control group.
Laminectomy time per spinal segment | Immediately after surgery.
  Laminectomy time for a single spinal segment = total laminectomy time ÷ Number of spinal segments with laminectomy.
Total laminectomy time | Immediately after surgery.
  The time from the start of laminectomy until the tool stops working is denoted as the total laminectomy time.
Operative time | Immediately after surgery.
  From the time the skin is cut to the time the suture is finished.
Amount of surgical bleeding | Immediately after surgery.
  Amount of surgical bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Weishi Li, M.D., Principal Investigator — Peking University Third Hospital
Locations (3):
- China (3):
  - Peking University Third Hospital, Beijing
  - Third Affiliated hospital of Southern medical university, Guangzhou
  - Zhejiang Provincial Hospital of Chinese Medicine, Hangzhou

IPD SHARING:
Plan to Share IPD: No